CLINICAL TRIAL: NCT06087653
Title: A Protocol to Assess the Safety, Efficacy, and Pharmacokinetics of Continuous Subcutaneous Administration of Low-dose Lenalidomide (STAR-LLD) for the Treatment of Multiple Myeloma (MM)
Brief Title: Safety, Efficacy, and Pharmacokinetics of Continuous Subcutaneous Lenalidomide in Multiple Myeloma (MM)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Starton Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAR LLD MM 023
Record Dates: First submitted 2023-09-20; First posted 2023-10-18 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Dose defining study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- ARM1 - Lenalidomide 400 mcg/h (Experimental): Lenalidomide 400 mcg/hr continuously for 28 of 28-day cycle
  Interventions: Drug: Lenalidomide
- Arm2 - Lenalidomide 300 mcg/h (Experimental): Lenalidomide 300 mcg/hr continuously for 28 of 28-day cycle
  Interventions: Drug: Lenalidomide
- Arm 3 - Lenalidomide 500 mcg/h (Experimental): Lenalidomide 500 mcg/hr continuously for 28 of 28-day cycle
  Interventions: Drug: Lenalidomide
- Arm 4 - Lenalidomide 600 mcg/h (Experimental): Lenalidomide 600 mcg/hr continuously for 28 of 28-day cycle
  Interventions: Drug: Lenalidomide
- Arm 5 - Lenalidomide oral capsule control (Active Comparator): Lenalidomide 25mg/d oral capsules continuously for 28 of 28-day cycle
  Interventions: Drug: Lenalidomide 25 MG Oral Capsule

INTERVENTIONS:
Drug: Lenalidomide — Low-dose lenalidomide continuous SC infusion (STAR-LDD) in combination with bortezomib and dexamethasone
  Other Names: bortezamib; dexamethasone
  Arms: ARM1 - Lenalidomide 400 mcg/h; Arm 3 - Lenalidomide 500 mcg/h; Arm 4 - Lenalidomide 600 mcg/h; Arm2 - Lenalidomide 300 mcg/h
Drug: Lenalidomide 25 MG Oral Capsule — Oral lenalidomide for active control
  Arms: Arm 5 - Lenalidomide oral capsule control

SUMMARY:
Primary Objective • Assess the safety and tolerability of low-dose lenalidomide administered by continuous subcutaneous (SC) infusion (STAR-LLD) in combination with dexamethasone and a proteasome inhibitor (PI).

Secondary Objectives

* • To establish the pharmacokinetic (PK) profile of STAR-LLD at a defined infusion rate targeting steady-state blood concentrations.
* • Evaluate changes in efficacy indicators including objective response rate (ORR), progression-free survival (PFS), and duration of response (DOR).

Exploratory Objective

* To assess the impact of STAR-LLD on patient reported symptoms and outcomes. Primary Endpoints
* The grade, frequency, and relationship of treatment-emergent adverse events (TEAEs) including adverse events of special interest (AESIs): (gastrointestinal [GI] toxicity, fatigue, hematologic toxicity, rash (non-infusion site).
* The observation of dose-limiting toxicities (DLTs) of STAR-LLD during Cycle 1. Secondary Endpoints

  •• Blood concentrations of lenalidomide at on Day 1 and at steady state.
* Changes in biomarkers during treatment.
* Rate of complete response, very good partial response (VGPR), partial response (PR), stable disease (SD), and progressive disease.
* Determination of ORR, PFS, and DOR

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years at the time of informed consent.
2. Autologous stem cell transplant (ASCT) ineligible.
3. SARS -CoV2 virus (COVID)-19 negative.
4. A prior diagnosis of MM as defined by International Myeloma Working Group (IMWG) criteria (Appendix 7).
5. Documented measurable disease following first line therapy defined as:

   * Serum monoclonal protein ≥1.0 g/dL by protein electrophoresis.
   * ≥200 mg/24 hours of monoclonal protein in the urine on 24-hour electrophoresis.
   * Serum free light chain (SFLC) ≥10 mg/dL AND abnormal serum kappa to lambda free light chain (FLC) ratio.
6. Intended to be treated in 2nd line or greater with lenalidomide, dexamethasone, and a PI.
7. Proteasome inhibitor sensitive defined as progression free for > 6 months from cessation of PI or never received a prior PI.
8. Progression per IMWG criteria on the most recent line of therapy.
9. Eastern Cooperative Oncology Group (ECOG-Appendix 1) performance status ≤2 (patients with a performance status of 3 based solely on bone pain secondary to MM may be eligible following consultation and approval by the Medical Monitor).
10. Willing to comply with the protocol defined Lenalidomide Pregnancy Risk Minimization Plan for the prevention of pregnancy (Appendix 5). Females of childbearing potential (FCBP) must have a medically supervised negative serum or urine pregnancy test 4-14 days prior to planned start of treatment and again 24 hours prior to initiation of study medication. All FCBP must agree to either commit to continued abstinence from sexual intercourse or begin TWO acceptable methods of birth control AT THE SAME TIME, at least 28 days before receiving the first dose of STAR-LLD. FCBP must also agree to ongoing pregnancy testing. Males must agree to use a latex or synthetic condom during sexual contact with a FCBP from the time of starting study treatment through 28 days after the last dose, even if they have had a vasectomy.
11. Able to take anti-thrombotic prophylaxis.
12. The following laboratory results must be met during screening:

    * ANC ≥1,000 cells/mm3 (1.0 x 109/L).
    * Platelet count ≥75,000 cells/mm3 (75 x 109/L).
    * Hemoglobin ≥8.0 g/dL (red blood cell (RBC) transfusions are permitted prior to initiation of study drug if hemoglobin is stable for 72 hours).
    * Total bilirubin ≤1.5 x upper limit of normal (ULN), or patient diagnosed with Gilberts syndrome with a total bilirubin <5.0 x ULN that has been reviewed and approved by the Medical Monitor.
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 x ULN.
    * Calculated creatinine clearance ≥60 mL/min. Appendix 4
    * Negative pregnancy test for FCBP (must be obtained within 4-14 days before the initiation of study drug.
13. The following criteria must be met within 72 hours prior to first administration of continuous infusion STAR-LLD:

    * ANC ≥1,000 cells/mm3 (1.0 x 109/L).
    * Platelet count ≥75,000 cells/mm3 (75 x 109/L).
    * Hemoglobin ≥8.0 g/dL (RBC transfusions are permitted prior to initiation of study drug if hemoglobin is stable for 72 hours).
    * Calculated creatinine clearance ≥60 mL/min. Appendix 4
    * Negative pregnancy test for FCBP (must be obtained within 24 hours of first dose of study drug).
14. Able and willing to receive percutaneous ambulatory therapy.
15. Has an in-home care partner willing to receive training from a nurse for assistance with pump management.

Exclusion Criteria:

1. Pregnant or breastfeeding.
2. Received an ASCT.
3. Venous thromboembolism within 12 months of starting treatment on study.
4. Patients with active hepatitis B or C or human immunodeficiency virus (HIV) positive and on active therapy for those viral illnesses.
5. Currently taking any investigational therapy for the treatment of MM. A 28-day washout prior to Cycle 1 Day 1 is required for any previous investigational therapy.
6. Received a prior treatment line containing lenalidomide and failed to achieve an objective response (CR, VGPR or PR).
7. Discontinued a prior line of treatment due to intolerability to lenalidomide.
8. Concomitant use of strong CYP3A inducers (see https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers#table3-3).
9. Concurrent clinically significant amyloidosis or plasma cell leukemia or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes).
10. Known active infection requiring systemic anti-infective treatment (prophylactic treatment is permitted).
11. Prior malignancies within the previous 3 years, other than previously treated squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix or breast or another malignancy that is considered cured with minimal risk of recurrence (e.g., very low and low risk prostate cancer in active surveillance).
12. Prior major surgical procedure or radiation therapy within 4 weeks of the initiation of STAR-LLD (this does not include limited course of radiation used for management of bone pain within 7 days of initiation of STAR-LLD).
13. Any other condition that precludes adequate understanding, cooperation, and compliance with study procedures or any condition that could pose a risk to the patient's safety, as per the Investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and tolerability of low-dose lenalidomide administered by continuous subcutaneous (SC) infusion (STAR-LLD) in combination with dexamethasone and a proteasome inhibitor (PI). | 12 months
  Based on the incidence of adverse events associated with the use of the drug

SECONDARY OUTCOMES:
To assess the immunologic activity of natural killer (NK) cells and T cells for innate and humoral immunity. | 12 months
  Measure changes in T cell and NK cell function/exhaustion over the study by flow cytometry
To establish the pharmacokinetic (PK) profile of STAR-LLD at a defined infusion rate targeting steady-state blood concentrations. | 12 months
  Meaured vs predicted blood concentrations of lenalidomide during the infusion and at steady state
To determine pharmacodynamic (PD) changes with STAR-LLD in a panel of biomarkers associated with clinical response to lenalidomide. | 12 months
  Evaluate desirable changes in immune cells activity over therapy
Evaluate changes in efficacy indicators including objective response rate (ORR), progression-free survival (PFS), and duration of response (DOR). | 12 months
  An ORR of 60% is representative of patients being retreated with PI and Len

OTHER OUTCOMES:
Assess the DOR, PFS during treatment | 18 months
  Report the deprived data for these outcomes

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Regional Oncology Center, Wilson, North Carolina
  - Gabrail Cancer & Research Center, Canton, Ohio

IPD SHARING:
Plan to Share IPD: No